CLINICAL TRIAL: NCT00282594
Title: No Outcome Benefit for the Use of Intensive Insulin Therapy in the Critically Ill General and Vascular Surgical Patient. A Randomized Prospective Trial.
Brief Title: The Effect of Intensive Insulin Therapy in the Surgical Critical Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genesys (Other)
Collaborators: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRMC 050023
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Last update posted 2006-01-27 (Estimated); Status verified 2005-11

CONDITIONS: Sepsis; Respiratory Failure; Renal Failure; Surgical Site Infection
Keywords: Intensive Insulin Therapy; General Surgical; Vascular Surgical; Tight Glycemic Control
MeSH Terms: conditions — Sepsis; Respiratory Insufficiency; Renal Insufficiency; Surgical Wound Infection | interventions — Insulin

INTERVENTIONS:
Drug: Novolin R (human recombinant Insulin)

SUMMARY:
We sought to determine if there is a benefit to using an insulin drip to control hyperglycemia in the surgical critical care unit for patients who undergo general and vascular surgery.

DETAILED DESCRIPTION:
While evidence exists for using tight glycemic control in the critically ill cardiac surgical patient, other patient populations have yet to be studied. We performed a prospective randomized trial for using intensive insulin therapy in the general and vascular critically ill surgical patient population. We will compare tight glycemic control versus conventional glycemic control to determine if there is a benefit to the normalization of blood glucose levels in this patient population

ELIGIBILITY:
Inclusion Criteria: Patients undergoing a general or vascular surgical procedure requiring admission to the surgical intensive care unit as a result of ventilatory requirement, vasopressor support, or physiologic instability

-

Exclusion Criteria:

* Under age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317
Dates: Start 2003-07; Study Completion 2005-10

PRIMARY OUTCOMES:
Mortality

SECONDARY OUTCOMES:
Length of ICU Stay
Ventilatory Requirement
Vasopressor Support
Incidence of Renal Failure
Incidence of Wound Infection

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kia, DO, Principal Investigator — Ascension Health
Locations (1):
- Genesys Regional Medical Center, Grand Blanc, Michigan, United States

REFERENCES:
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168